CLINICAL TRIAL: NCT00538876
Title: Phase I Study of Epigenetic Priming Using Decitabine With Induction Chemotherapy in Patients With Acute Myelogenous Leukemia (AML)
Brief Title: Phase I Epigenetic Priming Using Decitabine With Induction Chemotherapy in AML
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Joseph Scandura, MD, Weill Cornell Medical College
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0704009108
Record Dates: First submitted 2007-10-02; First posted 2007-10-03 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2011-06

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine

INTERVENTIONS:
Drug: decitabine — Decitabine will be administered by intravenous injection at a dose of 20 mg/m2/day as a daily 1hr infusion (Arm A) or by continuous infusion (Arm B) for 3, 5 or 7 days. On the day following the final dose of decitabine, standard "7+3" induction chemotherapy will begin.

SUMMARY:
This is an open label phase I study designed to explore the feasibility, safety and biologic activity of epigenetic priming with decitabine prior to standard cytarabine, daunorubicin induction chemotherapy in younger patients with less-than-favorable risk AML.

Primary Objective: To find an appropriate dose level for decitabine when used as priming for cytarabine and daunorubicin "7+3" induction chemotherapy in AML.

Secondary Objectives:

1. To establish the safety and expected toxicities of decitabine when used as priming for cytarabine and daunorubicin "7+3" induction chemotherapy in AML.
2. To establish the optimal dose schedule of decitabine required to broadly demethylate cytosine residues in genomic regulatory regions.
3. To investigate, in selected cases, the molecular and cellular consequences of decitabine-induced hypomethylation by a) establishing the extent and degree of hypomethylation at specific genomic loci required to reactivate the expression of repressed genes and by b) determining the effect of hypomethylation on the differentiation and/or apoptosis of leukemic blasts.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed diagnosis of Acute Myelogenous Leukemia (AML)
* Patient is >18 and ≤ 60 years of age.
* AML subgroup is associated with less-than-favorable risk as defined by:

  * The absence of good risk molecular features: t(8;21), inv(16), t(16;16), or t(15;17) translocations identified by FISH or standard metaphase karyotyping or evidence for the corresponding fusion transcripts, AML1-ETO, CBFβ-SMMHC, or PML-RARα, as identified by RT-PCR or suggested by the FAB M3 phenotype;
  * A history of an antecedent myelodysplastic syndrome;
  * A history of an antecedent Philadelphia-chromosome negative myeloproliferative disorder (e.g., polycythemia vera, essential thrombocythemia, primary myelofibrosis);
  * Treatment-related AML believed secondary to prior cytotoxic chemotherapy for an unrelated disease.
* Patient has adequate cardiac function as defined by:

  * An echocardiogram or MUGA scan demonstrating an ejection fraction within normal limits.
* ECOG performance status > = 2.
* Patient has adequate hepatic/renal function as defined by:

  * Total bilirubin ≤ 2 mg/dL. Patients with documented evidence of Gilbert's Syndrome resulting in elevated total bilirubin levels will be eligible, provided all other eligibility criteria are met.
  * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤1.5 x the ULN.
  * Creatinine ≤ 2 mg/dL (or a creatinine clearance >50 mL/min/1.73 m2, by direct measure).
* Patient is not childbearing:

  * Female subjects must be surgically sterile, postmenopausal, or have a β-HCG indicating that they are not pregnant at the time screening is performed.
  * Female patients of childbearing potential must agree to take appropriate measures to ensure that they do not become pregnant while enrolled on protocol (i.e., within 2 months of administration of chemotherapy).
  * Male patients must agree to take appropriate measures to ensure that they do not father a child while enrolled on protocol (i.e., within 2 months following administration of chemotherapy).
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* AML with "good risk" molecular features: karyotype demonstrating the presence of t(8;21), inv(16), t(16;16), or t(15;17) translocations identified by FISH or standard metaphase karyotyping or evidence for the corresponding fusion transcripts, AML1-ETO, CBFβ-SMMHC, or PML-RARα, as identified by RT-PCR or suggested by the FAB M3 phenotype.
* Patient has a history of chronic myelogenous leukemia or has molecular evidence of the t(9;22) translocation by FISH, metaphase karyotype or RT-PCR for the BCR-ABL fusion transcript.
* Patient has received chemotherapy (other than hydroxyurea) or radiation within the 2 weeks prior to planned therapy on this study.
* Patient has an active second malignancy.
* Patient has a medical condition or illness considered by the Investigator to constitute an unwarranted high risk for investigational drug treatment.
* Patient has an uncontrolled serious infection.
* Patient is pregnant or nursing an infant.
* Patient has a psychiatric disorder or altered mental status that would preclude understanding of the informed consent process and/or completion of the necessary studies.
* Patient has an inability or unwillingness, in the opinion of the Investigator, to comply with the protocol requirements.
* Patients with central nervous system (CNS) (or leptomeningeal) involvement by their AML may be considered for treatment at the Investigator's discretion and following discussion with the Medical Monitor, in order to allow for appropriate management.
* Patient has circulating blast count > 50,000/μL (patients may be enrolled if circulating blast count is controlled by hydroxyurea and/or, if clinically indicated, by leukopheresis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To establish the safety and expected toxicities of decitabine when used as priming for cytarabine and daunorubicin "7+3" induction chemotherapy in AML | duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Scandura, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States

REFERENCES:
- [Result] Scandura JM, Roboz GJ, Moh M, Morawa E, Brenet F, Bose JR, Villegas L, Gergis US, Mayer SA, Ippoliti CM, Curcio TJ, Ritchie EK, Feldman EJ. Phase 1 study of epigenetic priming with decitabine prior to standard induction chemotherapy for patients with AML. Blood. 2011 Aug 11;118(6):1472-80. doi: 10.1182/blood-2010-11-320093. Epub 2011 May 25. PMID 21613261